CLINICAL TRIAL: NCT04915365
Title: Effect of Acetazolamide on Right Heart Function at Rest in Lowlanders With Chronic Obstructive Pulmunary Disease (COPD) Traveling to High Altitude
Brief Title: Effect of Acetazolamide on Right Heart Function at Rest in Lowlanders With COPD Traveling to High Altitude
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine, Kyrgyz Republic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01-2021-SU-HAECHO
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Right Heart Function; Chronic Obstructive Pulmonary Disease; Altitude Sickness
Keywords: Acetazolamide; Mountain sickness; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Altitude Sickness; Hypertension, Pulmonary | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, double-blind
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) An independent pharmacist will prepare identically looking active and placebo capsules labelled with secret codes. Codes will be concealed to investigators and patients until completion of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide (oral capsules @125 mg), starting dose 3 capsules (375 mg), subsequent doses 1 capsule (125 mg) in the morning, 2 capsules (250 mg) in the evening, administered in qualifying participants, during the stay at 3100 m.
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo (oral capsules, identically looking as active drug), starting dose 3 capsules, subsequent doses
  1 capsule in the morning, 2 capsules in the evening, administered in qualifying participants, during the stay at 3100 m.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide (oral capsules @125 mg), starting dose 3 capsules (375 mg), subsequent doses 1 capsule (125 mg) in the morning, 2 capsules (250 mg) in the evening, administered in qualifying participants, during the stay at 3100 m.
  Other Names: Acetazolamide, oral capsule
  Arms: Acetazolamide
Drug: Placebo — Placebo (oral capsules, identically looking as active drug), starting dose 3 capsules, subsequent doses
  1 capsule in the morning, 2 capsules in the evening, administered in qualifying participants, during the stay at 3100 m.
  Other Names: Placebo, oral capsule
  Arms: Placebo

SUMMARY:
The purpose of this randomized, placebo-controlled double-blind trial is to evaluate the effect of acetazolamide on right heart function at rest in lowlanders with chronic obstructive pulmonary disease (COPD) traveling to high altitude (HA) and developing early signs of altitude-illness.

DETAILED DESCRIPTION:
This randomized placebo-controlled, double-blind, parallel-design trial will evaluate effect of acetazolamide on right heart function in lowlanders with chronic obstructive pulmonary disease (COPD) travelling to high altitude and developping early symptoms and/or signs of impending altitude-illness. Qualifying participants will be randomized 1:1 to acetazolamide or placebo treatment during their further stay of 2 days at 3'100 m.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 35-75 y, living at low altitude (<800 m).
* COPD diagnosed according to the Global Initiative for Obstructive Lung Disease (GOLD) guidelines, FEV1 40-80% predicted, pulse oximetry

  ≥92%, PaCO2 <6 kPa, breathing ambient air at 760 m.
* One of the following early signs and/or symptoms of impending altitudeillness identified by self-monitoring during ascent to or stay at 3100 m:
* Pulse oximetry SpO2≤84%
* Headache or nausea/vomiting or fatigue/weakness or dizziness/lightheadedness of at least moderate intensity

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia or hypercapnia at 760 m (see above).
* Other lung disease, relevant comorbidities (such as uncontrolled cardiovascular disease, i.e., unstable arterial hypertension, coronary artery disease; previous stroke; obesity (body mass index >35 kg/m2); internal, neurologic, rheumatologic or psychiatric disease; current heavy smoking (>20 cigarettes per day).
* Renal failure and/or allergy to sulfonamides.
* Patients who do not have early signs and/or signs of impending altitudeillness by self-monitoring (as defined above) at 3'100m will not be included.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change of pulmonary artery pressure | 3 days
  Difference in change of pulmonary artery pressure (RV/RA) evaluated by echocardiography at 3100 m in the acetazolamide compared to the placebo group

SECONDARY OUTCOMES:
Difference in change of pulmonary artery pressure (RV/RA) low altitude versus high altitude | 3 days
  Difference in change of pulmonary artery pressure evaluated by echocardiography from 760 m baseline measurement to measurement at 3100 m in the acetazolamide compared to the placebo group
Difference in cardiac output | 3 days
  Difference in change of cardiac output evaluated by echocardiography in the acetazolamide compared to the placebo group
Difference in right heart dimensions | 3 days
  Difference in change of right heart dimensions evaluated by echocardiography in the acetazolamide compared to the placebo group
Difference in right heart function | 3 days
  Difference in change of tricuspid annular plane systolic sxcursion (TAPSE) evaluated by echocardiography in the acetazolamide compared to the placebo group
Difference in right heart function | 3 days
  Difference in change of fraction area change (FAC) evaluated by echocardiography in the acetazolamide compared to the placebo group
Difference in right heart function | 3 days
  Difference in change of tissue dopple S (TDI S) evaluated by echocardiography in the acetazolamide compared to the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof, Study Chair — University Hospital, Zürich, Switzerland; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No